CLINICAL TRIAL: NCT02810158
Title: Diagnosis of Obstructive Sleep Apnoea by Selective Secondary Electrospray Ionization - Mass Spectrometry (SESIMS)
Brief Title: Mass Spectral Fingerprinting in Obstructive Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC-Nr.2016-00384
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Obstructive Sleep Apnoea (OSA); Exhaled Breath; Mass Spectrometry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with suspected OSA: Persons with clinical suspicion of obstructive sleep apnoea syndrome (OSA)

SUMMARY:
To answer the question whether a previously detected breath profile in patients suffering from obstructive sleep apnoea (OSA) can be found in a cohort of patients with suspected OSA using mass spectrometry (validation study).

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of obstructive sleep apnoea syndrome (based on clinical symptoms such as increased daytime sleepiness; Epworth Sleepiness Score (ESS) > 10).
* Age between 18 and 85 years at study entry.

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of OSA
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
OSA-specific mass spectrometric pattern of VOCs in the exhaled breath | one hour, single measurement, no follow-up
  Concentration of volatile organic compounds (VOCs) in the exhaled breath will be analysed using mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof. MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Nowak N, Engler A, Thiel S, Stoberl AS, Sinues P, Zenobi R, Kohler M. Validation of breath biomarkers for obstructive sleep apnea. Sleep Med. 2021 Sep;85:75-86. doi: 10.1016/j.sleep.2021.06.040. Epub 2021 Jul 3. PMID 34280868